CLINICAL TRIAL: NCT02706639
Title: Williams Syndrome (WS) and Supravalvar Aortic Stenosis (SVAS) DNA and Tissue Bank
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160074; 16-H-0074
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09-16

CONDITIONS: Williams Syndrome; Supravalvular Aortic Stenosis; Cardiovascular Disease
Keywords: Biospecimen Procurement; Laboratory Research Specimens; Sample Collection; Rare Diseases; Natural History
MeSH Terms: conditions — Williams Syndrome; Aortic Stenosis, Supravalvular; Cardiovascular Diseases; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- SVAS/SVAS-like group: Children or adults must: be between the ages of 0-85; have clinical features of SVAS; SVAS-like condition; have genetic testing results that imply affected status (SVAS has decreased penetrance)
- Unaffected related (family member) controls: Children or adults: family members be between the ages of one month old and 85 years old, not carry a diagnosis of WS, SVAS, an SVAS-like condition or a known (at the time of enrollment) WS gene region variant.
- Unaffected unrelated controls: Adults, 18-85: unrelated controls be between the ages 18 and 85 years old, not carry a diagnosis of WS, SVAS, an SVAS-like condition or a known (at the time of enrollment) WS gene region variant.
- WS group: Children or adults must: be between the ages of 0 and 85; have a presumed or confirmed diagnosis of WS; have a parent/guardian available to provide consent and assist in answering medical questions
- WS region gene changes: Children or adults must: be between the ages of 0-85; have clinical or research genetic testing that reports gene variation in one or more genes in the WS region (ELN variants alone will be considered in the SVAS category but other changes to the region that include ELN plus other genes may be grouped in this category).

SUMMARY:
Williams syndrome is a rare genetic disorder occurring in 1:8000-12,000 individuals. It is caused by the deletion of 25-27 coding genes, including elastin (ELN) on the 7th human chromosome. Haploinsufficiency for these genes leads to the features of the condition, including:

* Distinctive facial features;
* Characteristic vascular problems including hypertension, focal vascular stenosis, (when present in the aorta this is referred to as SVAS), vascular stiffness and differences in heart rate variability;
* Endocrine abnormalities including hypercalcemia, hypothyroidism, and early puberty;
* Metabolic concerns with colic and failure to gain weight in infancy and obesity and early glucose intolerance in adulthood;
* Characteristic neurocognitive profile comprised of cognitive impairment, high sociality with concurrent social awkwardness, difficulty with visual-spatial tasks, relative strengths in speech, and lack of social fear;
* Anxiety and chronic pain in adulthood

Most individuals with WS carry the same basic deletion on Chromosome 7q11.23. However, each feature may present as mild or more severe in any given individual. Variation in the presence and severity of these vascular phenotypes remains unexplained.

The supravalvar aortic stenosis (SVAS) phenotype is caused by haploinsufficiency for elastin. This can come about due to the WS deletion (as above) or due to heterozygous variation in elastin (ELN) gene itself in this region. When this protein is reduced, connective tissues lose its strength, flexibility, and overall support. When this happens in the aorta, it may cause vascular narrowing that presents as shortness of breath, chest pain, and even heart failure if left untreated. Narrowing also occurs in other vessels especially the pulmonary and renal arteries. Changes in non-vascular elastic tissues such as the skin and lungs also occur. As in WBS, phenotypic variation also occurs in people with ELN gene changes--This variability remains unexplained despite all the on-going research.

Most individuals with features of SVAS have either WS or an elastin variant. There are, however, a smaller number of individuals with the phenotypic features of the condition whose genetic underpinnings are yet to be defined (they are referred to as SVAS-like).

Additionally, there are 26 other coding genes within the WS critical region that contribute to various other features of the condition

Objective:

1. To collect historical information and to bank DNA, cells, and tissue from individuals with genetic alterations in the WS/ELN gene region, those with an SVAS -like phenotype and unaffected family members/controls to facilitate future research into the many phenotypes seen in these individuals.
2. Currently, we plan to use the collected samples to identify genetic and environmental factors that contribute to the variability in different phenotypes (vascular and non-vascular) in individuals with WS, SVAS and SVAS-like conditions, individuals with variation in WS genes other than elastin and unaffected family members and controls. For the non-vascular features of WS and SVAS-like conditions for which a specific gene has not been implicated in the disease, we would also like to identify causative genes as well as modifiers. Likewise, by evaluating people with variation in other WS region genes, we can determine what contribution those genes make to the studied phenotypes. Controls will be both used to assess the frequency of genetic features in people without the phenotype in question and to evaluate heritability, penetrance, and expressivity of relevant variants.

Eligibility:

People ages 0-85 with either WS, SVAS, and/or an SVAS-like condition, unaffected family members or adult unrelated controls.

Design:

This study is not a treatment protocol.

This study will consist of:

Collection of personal history (questionnaires) and medical record data (relevant physician notes, lab and diagnostic tests and studies) to study the natural history of these conditions, allow stratification of disease severity, and identification of environmental risk factors;

Collection of blood, saliva, urine and surgical tissue waste to allow DNA and RNA preparation as well as study of tissues both in situ and through the generation of IPSCs;

Expression studies on available tissues (lymphocytes, IPSCs, vascular, skin, other collected tissues) to look for differential regulation of target genes;

Direct imaging of tissues (lymphocytes, IPSCs, vascular, skin, other collected tissues);

Storage of collected data and specimens for future research;

A questionnaire may be sent to participants or parent/guardian or LAR to respond on behalf of participant.

DETAILED DESCRIPTION:
Our goal with the Williams syndrome (WS) and Supravalvar Aortic Stenosis (SVAS), deoxyribonucleic acid (DNA) and Tissue Bank is to collect enough samples from individuals with these rare conditions to ask questions about the genes that cause the many WS and SVAS related phenotypes, and to determine the genetic and environmental changes that modify the severity of disease from person to person. In addition, we would like to learn more about the natural history of these conditions and if there are environmental or genetic signatures that are associated with symptom presence.

The protocol detailed here will provide for the collection of historical information, laboratory and imaging data, DNA and tissue to perform these studies now and in the future. Because technology changes rapidly and because this is a rare condition, our goal is to generate a collection that will be available for analysis for many years.

In addition to DNA and tissue collection proposed, we would like to begin to use the specimens collected here to continue to ask questions about genetic changes within and outside of the WS critical region that influence disease outcomes, including primary disease drivers and modifiers of disease severity. Our primary focus is on drivers of vascular disease in WS, WS-region variation, SVAS and SVAS-like conditions, but investigation of genetic and environmental factors that influence other systems is also anticipated.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will recruit individuals with WS, SVAS or SVAS-like conditions, individuals with variation in WS genes other than ELN and unaffected family members or unrelated controls

Children or adults participating in this study as part of the WS group must:

* be between the ages of 0 and 85
* have a presumed or confirmed diagnosis of WS (typical or atypical deletions overlapping the WS region are acceptable, as are clinical diagnoses made by a physician familiar with WS) have a parent/guardian available to provide consent and assist in answering medical questions

Children or adults participating in the study as part of the SVAS/SVAS-like group must:

* be between the ages of 0 and 85
* have clinical features suggestive of SVAS or an SVAS-like condition OR have no clinical features of SVAS or of an SVAS-like condition but have genetic testing results that imply affected status (SVAS has decreased penetrance).

Have a parent/guardian available to provide consent and assist in answering medical questions if they are a minor (not applicable to adults)

Children or adults with WS region gene changes (variation affecting one or more WS region genes):

* be between the ages of 0 and 85
* have clinical or research genetic testing that reports gene variation in one or more genes in the WS region (ELN variants alone will be considered in the SVAS category but other changes to the region that include ELN plus other genes may be grouped in this category).

Have a parent/guardian available to provide consent and assist in answering medical questions if they are a minor or if they have cognitive impairment that would impede their ability to consent on their own behalf.

Children or adults serving as unaffected family members or adult unrelated controls must:

* family members be between the ages of one month old and 85 years old
* unrelated controls be between the ages 18 and 85 years old
* not carry a diagnosis of WS, SVAS, an SVAS-like condition or a known (at the time of enrollment) WS gene region variant.
* In some cases, an individual may appear to be unaffected, but upon genetic testing may be found to be an asymptomatic carrier for gene variant. If that happens, they will be transferred to the appropriate affected research group.

The eligible age range for unaffected family members participating in this study includes all family members from one month onwards. This inclusive approach is undertaken to comprehensively grasp the affected status across all family members, avoiding any form of age-based discrimination. Understanding that certain cases may not exhibit phenotypic indications of affected status at a young age, it becomes crucial to gather early health characteristics of individuals who may initially appear unaffected but later manifest disease findings. Participation in research, as previously noted, has a potential to identify people at risk who were previously thought to be healthy.

Ages: 1 Day to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Affected: 1) people with WS (adults and children), 2) people with ELN-related SVAS (adults and children), 3) people with SVAS-like conditions (those with an SVAS phenotype but no known pathologic variant in ELN, (adults and children)) 4) individuals with single or oligogenic variation in WS genes other than ELN (adults and children) Unaffected: 5) unaffected family members of participating subjects (children or adults), enrolled as controls 6) unrelated unaffected adult controls.
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2040-09-25 (Estimated); Study Completion 2040-09-25 (Estimated)

PRIMARY OUTCOMES:
To collect historical information and bank specimens form individuals with Williams Syndrome and SVAS for future research | ongoing
  The overall objective of this study is to collect historical information and to bank DNA, cells and tissue from individuals with WS and SVAS to facilitate future research into the many phenotypes seen in these individuals.

SECONDARY OUTCOMES:
To identify genetic and environmental factors that contribute to the variability in different phenotypes in individuals with WS, SVAS, and SVAS-like conditions | ongoing
  To identify genetic and environmental factors that contribute to the variability in different phenotypes (vascular and non-vascular) in individuals with WS, SVAS and SVAS-like conditions. For the non-vascular features of WS and SVAS-like conditions for which a specific gene has not been implicated in the disease, we would also like to identify causative genes.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Boehm, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-H-0074.html